CLINICAL TRIAL: NCT01606501
Title: Outcomes Following Severe Distal Tibia, Ankle and/or Foot Trauma: Comparison of Limb Salvage Versus Transtibial Amputation Protocol (OUTLET Study)
Brief Title: Outcomes Following Severe Distal Tibia, Ankle and/or Foot Trauma: Comparison of Limb Salvage Versus Transtibial Amputation Protocol
Acronym: OUTLET
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWH-09-2-0108-OUT
Record Dates: First submitted 2012-04-16; First posted 2012-05-25 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Severe Distal Tibia Injury; Severe Ankle Injury; Severe Foot Injury; Major Soft Tissue Loss; Major Bone Articular Surface Loss; Major Ankle Articular Surface Loss
MeSH Terms: conditions — Ankle Injuries; Foot Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Limb Salvage patients: Patients undergoing limb salvage following severe distal tibia, ankle and/or foot injuries with major soft tissue, bone and/or ankle articular surface loss.
- Transtibial Amputation patients: Patients undergoing transtibial amputation following severe distal tibia, ankle and/or foot injuries with major soft tissue, bone and/or ankle articular surface loss.

SUMMARY:
The primary aim this prospective longitudinal observational outcomes study is to compare 18 month functional outcomes and health related quality of life (HRQoL) of patients undergoing salvage versus amputation following severe distal tibia, ankle and/or foot fractures with major soft tissue, bone and/or ankle articular surface loss. Functional outcomes and HRQoL will be measured using well established self reported measures, including the Veterans Rand Health Survey (VR-12) and the Short Musculoskeletal Functional Assessment (SMFA).

Hypothesis 1: As a group, salvage patients with severe distal tibia, ankle and/or foot injuries with major soft tissue, bone and/or ankle articular surface loss will have similar functional outcomes and HRQoL had they undergone a transtibial amputation (within 6 weeks of injury).

Hypothesis 2: The subgroup of salvage patients who have either (1) a soft tissue injury that requires tissue transfer; (2) articular damage requiring arthrodesis of the ankle joint; or (3) bone loss at the distal tibia or ankle will have better functional outcomes and HRQoL had they undergone a transtibial amputation (within 6 weeks of injury).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an injury that meets at least one of the following:

   1. Gustilo type III pilon fractures consistent with one of the following OTA codes: 43B1.3, 43B2-B3, 43C, 44B, 44C
   2. Gustilo type III B or C ankle fractures
   3. Gustilo type III mid and/or hind foot fractures consistent with one of the following OTA codes: 81B2-B3, 82B and 82C
   4. Open foot crush or blast injuries from high energy mechanism involving the mid and /or hind foot with significant soft tissues damage
   5. Other severe foot injury (including closed foot crush or blast injuries)
2. Ages 18-60 inclusive.
3. Admitted to the hospital prior to definitive wound closure.

Inclusion notes:

1. Patients may have other injuries except as noted below under exclusion criteria.
2. Foot crush and blast injuries are eligible if they are considered to be at significant risk for impaired outcome with moderate to severe disability and typically include one of the following associated injuries:

   1. ankle dislocation (80A)
   2. subtalar dislocation (80B)
   3. extruded talus
   4. chopart dislocation (80C)
   5. multiple midfoot dislocations (80C)
   6. three or greater proximal metatarsal fractures
   7. heel pad/plantar degloving
   8. extensive muscle necrosis in an open injury from crush, ischemia and/or foot compartment syndrome
3. These injuries may include "toe-pan" injuries from motor vehicle accidents and crush-like injuries from motorcycle accidents, and traumatic amputations.

Exclusion Criteria:

1. Patient has a Glasgow Coma Scale motor score of 0-4 or a Glasgow Coma Scale motor score of 5 with a significant traumatic brain injury (defined as an AIS code of 5 or 6) at time of consent
2. Patient has third degree burns on >10% total surface area affecting the study limb
3. Patient has a previous leg or foot amputation of either limb
4. Patient is non-ambulatory due to an associated complete spinal cord injury
5. Patient non-ambulatory pre-injury
6. Patient speaks neither English nor Spanish
7. Patient likely to have severe problems with maintaining follow- up due to at least one of the following:

   1. Patient has been diagnosed with a severe psychiatric condition
   2. Patient is intellectually challenged without adequate family support
   3. Patient lives outside the hospital's catchment area
   4. Follow-up is planned at another medical center
   5. Patients who are prisoners or homeless

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be patients aged 18-60 with severe open or crushed distal tibia, ankle and/or foot injury that go on to limb salvage or receive a below the knee amputation.
Sampling Method: Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2012-05; Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Patient reported function and health related quality of life | 18 months
  Functional Outcomes and health related quality of life will be measured using well established self reported measures, including the Veterans RAND Health Survey (VR-12) and the Short Musculoskeletal Functional Assessment (SMFA).

SECONDARY OUTCOMES:
Physical impairment | 18 months
  Physical impairment will be determined using objective performance measures of agility (4 step square test and Illinois Agility Test), strength and power (sit-to-stand test and timed stair climb), speed (self-selected walking speed and 40 yard shuttle run), postural stability (single leg stance) and overall activity will be measured using the step watch activity monitor.
Levels of participation | 18 months
  Levels of participation will be measured using self reported measures of return to usual major activity (work, active duty, school, home management) and the Paffenbarger Activity Scale (PPAQ) that measures participation in light, moderate and vigorous recreational or sports activities.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bosse, MD, Principal Investigator — Carolinas Medical Center; Lisa Reider, MHS, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Navy Medical Center San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Walter Reed National Military Medical Center, Washington D.C., District of Columbia
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Florida Orthopaedic Institute, St. Joseph's Hospital, Tampa, Florida
  - Florida Orthopaedic Institute, Tampa General Hospital, Tampa, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - OrthoIndy Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa Medical Center, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth, Cleveland, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island/ Brown University, Providence, Rhode Island
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington/Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] McLaughlin KH, Mitchell SL, Archer KR, Master H, Morshed S, Gary JL, Jones CB, MacKenzie EJ, Reider L; METRC. Effect of Severe Distal Tibia, Ankle, and Mid- to Hindfoot Trauma on Meeting Physical Activity Guidelines 18 Months After Injury. Arch Phys Med Rehabil. 2022 Mar;103(3):409-417.e2. doi: 10.1016/j.apmr.2021.07.805. Epub 2021 Aug 21. PMID 34425087